CLINICAL TRIAL: NCT05247658
Title: Study Comparing a Therapeutic Lens Used Alone to a Therapeutic Lens Used in Association With an Amniotic Membrane Treated by the AMTRIX Process in Postoperative Care After Photorefractive Keratectomy (PRK)
Brief Title: Use of a Disk of Amniotic Membrane (Visio-AMTRIX) in Postoperative Care After PKR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of apparent benefits
Sponsor: TBF Genie Tissulaire (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AMTRIX-PKR-TBF; 2021-A01933-38 (Other: IDRCB)
Record Dates: First submitted 2022-02-09; First posted 2022-02-21 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Myopia; Astigmatism; Hypermetropia
Keywords: PhotoRefractive Keratectomy (PRK)
MeSH Terms: conditions — Myopia; Astigmatism; Hyperopia

STUDY DESIGN:
Intervention Model Description: Self-controlled trial: each patient serves as his or her own control. After bilateral PRK procedure, patients will receive both treatments, one treatment in each eye.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic lens alone (Active Comparator)
  Interventions: Other: Therapeutic lens alone
- Therapeutic lens + amniotic membrane (Visio-AMTRIX) (Experimental)
  Interventions: Other: Therapeutic lens + amniotic membrane (Visio-AMTRIX)

INTERVENTIONS:
Other: Therapeutic lens alone — Therapeutic lens will be apposed on patient's dominant eye after bilateral PRK. Therapeutic lens will be maintained without interruption until the first postoperative visit when it will be removed by the surgeon.
  Arms: Therapeutic lens alone
Other: Therapeutic lens + amniotic membrane (Visio-AMTRIX) — Amniotic membrane (Visio-AMTRIX) will be apposed under therapeutic lens on patient's non-dominant eye after bilateral PRK. Amniotic membrane and therapeutic lens will be maintained without interruption until the first postoperative visit when it will be removed by the surgeon.
  Arms: Therapeutic lens + amniotic membrane (Visio-AMTRIX)

SUMMARY:
The purpose of this open controlled multicenter trial is to assess the impact of use of an amniotic membrane on post PKR recovery.

DETAILED DESCRIPTION:
Photorefractive keratectomy (PRK) and laser-assisted in situ keratomileusis (LASIK) are two of the most widely used techniques of laser vision correction. However, one of the major disadvantages of the PRK technique is the pain experienced during 1 to 3 days after intervention.

Preliminary data on a limited number of patients tend to show a reduction of pain, tearing and discomfort in patients for whom a amniotic membrane was used under a therapeutic lens.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 80 years.
* Patient undergoing bilateral PRK procedure for myopia, astigmatism or hypermetropia with technique chosen for one of the following reasons: thin cornea, irregular cornea, suspected keratoconus, practice of combat or contact sports, professional activity at risk of direct impact.
* Patient understanding french language.
* Patient who received the study information and provided written consent to participation in the study.
* Patient who is a member or a beneficiary of a national health insurance plan.

Exclusion Criteria:

* Pregnant woman.
* Patient with a contraindication to PRK.
* Diabetic patient.
* Patient allergic to Oxybuprocaine and / or Tetracaine eye drops, to local anesthetics or to fluorescein.
* Monophthalmic patient.
* Person deprived of liberty by a judicial or administrative decision.
* Adult subjected to a legal protection measure or unable to express his / her consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
Change of pain in the eye treated with therapeutic lens + amniotic membrane (experimental) compared to eye treated with therapeutic lens alone (active comparator) | Day 1
  Pain evaluated from 0: no pain to 10: worst imaginable pain on visual analog scale (VAS) in both eyes

SECONDARY OUTCOMES:
Change of pain in the eye treated with therapeutic lens + amniotic membrane (experimental) compared to eye treated with therapeutic lens alone (active comparator) | 2 days, 3 days, 30 to 45 days
  Pain evaluated from 0: no pain to 10: worst imaginable pain on visual analog scale (VAS) in both eyes
Change of visual discomfort in the eye treated with therapeutic lens + amniotic membrane (experimental) compared to eye treated with therapeutic lens alone (active comparator) | 1 day, 2 days, 3 days, 30 to 45 days
  Evaluation by the patient of visual discomfort criteria; tearing, foreign body sensation, blurred vision, and photophobia; from 0: no discomfort to 10: worst imaginable discomfort on visual analog scale (VAS) in both eyes
Identical healing of both eyes | 2 or 3 days, 30 to 45 days
  Healing evaluated under slit lamp by fluorescein examination with measurement of ulcer size
Better visual acuity in the eye treated with therapeutic lens + amniotic membrane (experimental) compared to eye treated with therapeutic lens alone (active comparator) | 30 to 45 days
  Determination of logMAR values of uncorrected visual acuity and best corrected visual acuity for both eyes
Rate of corneal haze for each treatment | 30 to 45 days
  Evaluation of presence of corneal haze through the Hanna's grading scale from grade 0: no haze to grade 4: very severe haze

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Clinique Vision Laser des Alpes, Grenoble
  - Centre Monticelli-Paradis d'Ophtalmologie, Marseille
  - CHU de Saint-Etienne Hôpital Nord, Saint-Priest-en-Jarez